CLINICAL TRIAL: NCT03396874
Title: Gallium-68 PSMA-11 PET in Patients With Biochemical Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Morand Piert, MD, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM125841
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Cancer Metastatic; Prostate Cancer Recurrent
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patient participants (Experimental): PET/CT imaging
  Interventions: Drug: 68Ga-PSMA

INTERVENTIONS:
Drug: 68Ga-PSMA — PET/CT imaging with 68Ga-PSMA:
  68Ga-PSMA is an investigational radioactive drug that binds to receptors on prostate cancer cells. The intravenously administered drug dose will be about 5 mCi (range 3-7 mCi).
  Other Names: Gallium-68 PSMA-HBED-CC; Gallium-68 PSMA-11

SUMMARY:
This study evaluates the value of Gallium-68 labeled PSMA (68Ga-PSMA) for PET/CT imaging of prostate cancer recurrence. 68Ga-PSMA is a radioactive molecule, which binds to prostate cancer cells. Together with a PET/CT scanner, the distribution of 68Ga-PSMA can be determined in the body.

To test this new drug, participants will receive an intravenous injection of Ga-68-PSMA and then have a PET/CT scan. The scan results will be made available to study participants and treating physicians.

DETAILED DESCRIPTION:
This study evaluates Gallium-68 labelled PSMA-11 (also called Gallium-68 labelled PSMA-HBED-CC, or Gallium-68 labelled PSMA N,N'-bis(2-hydroxybenzyl)ethylenediamine-N,N'-diacetic acid), abbreviated here as 68Ga-PSMA. This molecule (or radiotracer) binds to receptors that are often present on prostate cancer cells. Using 68Ga-PSMA together with a positron emission tomography (PET) scanner (with computed tomography, called PET/CT), it is therefore possible to find prostate cancer lesions in the body. The study will test whether 68Ga-PSMA will identify prostate cancer more precisely than normal imaging methods (for example CT, MRI, or bone scan). A more precise identification of the location of the disease is important. Knowing where the disease is located will help to decide on the best course of action to treat the disease.

Men who have elevated tumor markers of prostate cancer are eligible for this study. Participants undergo a 68Ga-PSMA PET/CT scan before further treatment. Based on clinical information, including any prior imaging and biopsy/surgery information and follow-up information, we will determine whether 68Ga-PSMA PET/CT imaging was more accurate than the standard imaging. The study team will collect this information for up to 1 year after the 68Ga-PSMA PET/CT scan.

The results of the 68Ga-PSMA PET/CT scan will be shared with the participating patients. Also, results will be entered into the participant's medical record and shared with the treating physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological proven prostate adenocarcinoma.
2. Rising prostate specific antigen (PSA) after definitive therapy with prostatectomy or radiation therapy (external beam or brachytherapy).

   1. Post radical prostatectomy (RP) - according to American Urological Association (AUA) recommendation criteria: PSA greater than 0.2 ng/mL measured more than 6 weeks after RP and confirmatory persistent PSA greater than 0.2 ng/mL.
   2. Post-radiation therapy - according to ASTRO-Phoenix consensus definition: Nadir + greater than or equal to 2 ng/mL rise in PSA.
3. Karnofsky performance status of ≥ 50.
4. Age ≥ 18.
5. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Current investigational therapy for prostate cancer.
2. Unable to lie flat, still or tolerate a PET/CT scan.
3. Prior history of a malignancy within the last 2 years, except skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized, and except superficial bladder cancer.
4. Prisoner.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1435 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morand R Piert, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Codified data will be archived and stored in an imaging repository with limited metadata for analysis. Individuals seeking use of these data should contact the study chair. A data sharing contract for a HIPAA limited dataset will need to be executed prior to data sharing.
Supporting Information: CSR
Time Frame: Available as requested. Data will be archived indefinitely for research purposes.
Access Criteria: Individuals seeking use of these data should contact the study chair.

REFERENCES:
- [Result] Abghari-Gerst M, Armstrong WR, Nguyen K, Calais J, Czernin J, Lin D, Jariwala N, Rodnick M, Hope TA, Hearn J, Montgomery JS, Alva A, Reichert ZR, Spratt DE, Johnson TD, Scott PJH, Piert M. A Comprehensive Assessment of 68Ga-PSMA-11 PET in Biochemically Recurrent Prostate Cancer: Results from a Prospective Multicenter Study on 2,005 Patients. J Nucl Med. 2022 Apr;63(4):567-572. doi: 10.2967/jnumed.121.262412. Epub 2021 Jul 29. PMID 34326126

RESULTS

PARTICIPANT FLOW:
Groups:
- 68Ga-PSMA: Participants in this arm were prostate cancer patients who experienced elevated PSA after definitive therapy with prostatectomy, radiation therapy (external beam or brachytherapy), or focal therapy of the prostate.
- Physicians: Participants were the ordering physicians/practitioners of the patient participants in the 68Ga-PSMA study arm.
Period: Overall Study
Arm/Group | 68Ga-PSMA | Physicians
Started | 1181 | 254
68Ga-PSMA Scan | 1181 (received 68Ga-PSMA scan) | 0 (did not receive scans)
Completed | 1181 | 254
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 68Ga-PSMA | Physicians | Total
Number analyzed (Participants) | 1181 | 254 | 1435
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data not collected for the Physicians Arm
  years
    Age: number analyzed (Participants) | 1181 | 0 | 1181
    Age | 69.4 (7.0) |  | 69.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex: all male given disease (prostate cancer participants). Sex data not collected for the Physicians Arm.
  Participants
    number analyzed (Participants) | 1181 | 0 | 1181
    Female | 0 | 0 | 0
    Male | 1181 | 0 | 1181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data not collected for the Physicians Arm
  Participants
    number analyzed (Participants) | 1181 | 0 | 1181
    Hispanic or Latino | 6 |  | 6
    Not Hispanic or Latino | 1175 |  | 1175
    Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data not collected for the Physicians Arm
  Participants
    number analyzed (Participants) | 1181 | 0 | 1181
    American Indian or Alaska Native | 0 |  | 0
    Asian | 7 |  | 7
    Native Hawaiian or Other Pacific Islander | 0 |  | 0
    Black or African American | 99 |  | 99
    White | 1060 |  | 1060
    More than one race | 14 |  | 14
    Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1181 | 254 | 1435
Weight [Mean (Standard Deviation); unit: kg] — Population: Weight data not collected for the Physicians Arm
  kg
    number analyzed (Participants) | 1181 | 0 | 1181
    (all) | 91.2 (17.3) |  | 91.2 (17.3)
Height [Mean (Standard Deviation); unit: cm] — Population: Height data not collected for the Physicians Arm
  cm
    number analyzed (Participants) | 1181 | 0 | 1181
    (all) | 177.5 (8.7) |  | 177.5 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Positive Predictive Value (PPV) of 68Ga PSMA PET/CT for Detecting Prostate Cancer on a Per-patient Basis Confirmed by Histopathology.
Description: Evaluation of the positive predictive value (PPV) (true positives / (true positives + false positives)) of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by histopathology on a per-patient basis. On a per-patient basis, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%.
  The result of a histopathological examination of a PSMA positive lesion is obtained when available. Such data are collected as a single time point up to 12 months following the scan.
Time Frame: Up to 12 months after 68Ga-PSMA scan
Population: The participants analyzed were all those who had histopathological confirmation. Participants in this arm were prostate cancer patients who experienced elevated PSA after definitive therapy with prostatectomy, radiation therapy (external beam or brachytherapy), or focal therapy of the prostate.
Measure: Number (95% Confidence Interval); unit: percentage of times value is true
Groups:
- 68Ga-PSMA: PET/CT imaging
  68Ga-PSMA: PET/CT imaging with 68Ga-PSMA: 68Ga-PSMA is an investigational radioactive drug that binds to receptors on prostate cancer cells. The intravenously administered drug dose will be about 5 mCi (range 3-7 mCi).
Arm/Group | 68Ga-PSMA
Number analyzed (Participants) | 151
percentage of times value is true | 87.3 [81.58 to 100.00]
Statistical Analysis 1: Comparison: 68Ga-PSMA; We determined the positive predictive value (PPV) (true positives / (true positives + false positives)) of 68Ga-PSMA-11 PET for presence or absence of prostate cancer confirmed by histopathology on a per-patient basis. On a per-patient basis, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — The exact p-value cannot be entered as it is equal to 2.2e-16; Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); PPV = 87.3, 95% CI 2-sided [81.58 to 100.00]

2. Secondary Outcome: Sensitivity and PPV on a Per-patient and Per-region-basis of 68Ga-PSMA PET/CT for Detection of Tumor Location.
Description: The sensitivity and PPV of 68Ga-PSMA PET/CT is determined on a per-patient and per-region-basis for the detection of tumor location. Confirmation is obtained by conventional imaging, clinical follow-up, and/or histopathology/biopsy where available. Results of conventional imaging, clinical follow-up, and/or histopathology is collected as a single time point up to 12 months following the scan.
Time Frame: Up to 12 months after 68Ga-PSMA scan
Population: Participants analyzed were all those where either conventional imaging, clinical follow-up, or histopathology was available. Participants in this arm were prostate cancer patients who experienced elevated PSA after definitive therapy with prostatectomy, radiation therapy (external beam or brachytherapy), or focal therapy of the prostate.
Measure: Number (95% Confidence Interval); unit: percentage of times value is true
Arm/Group | 68Ga-PSMA
Number analyzed (Participants) | 516
percentage of times value is true
  PPV, Per-Participant Basis | 92.3 [90.0 to 100]
  Sensitivity, Per-Participant Basis | 95.29 [93.3 to 100.00]
  PPV, prostate or prostate bed | 91.1 [86.2 to 100.00]
  Sensitivity, prostate or prostate bed | 91.72 [86.74 to 100.00]
  PPV, pelvic lymph nodes | 90.78 [85.74 to 100.00]
  Sensitivity, pelvic lymph nodes | 96.97 [93.20 to 100.00]
  PPV, soft tissues | 91.25 [84.19 to 100.00]
  Sensitivity, soft tissues | 93.59 [86.99 to 100.00]
  PPV, bone | 95.17 [91.12 to 100.00]
  Sensitivity, bone | 100 [97.85 to 100.00]
Statistical Analysis 1: Comparison: 68Ga-PSMA; PPV, composite standard, per-patient basis: We determined the positive predictive value (PPV) of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy where available. On a per-patient basis, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, binomial proportion test — Per patient basis p-value = 2.2e-16; Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); PPV = 92.3, 95% CI 2-sided [90.0 to 100]
Statistical Analysis 2: Comparison: 68Ga-PSMA; Sensitivity, composite standard, per-patient basis: We determined the sensitivity of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy (composite standard of truth). On a per-patient basis, the sensitivity of conventional imaging ranges between 30-50%. The null hypothesis is that the sensitivity at 50% will be tested against the alternative hypothesis that the sensitivity is greater than 50%; Test type: Other — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Sensitivity — Per patient basis p-value = 2.2e-16; Sensitivity = 95.29, 95% CI 2-sided [93.3 to 100.00]
Statistical Analysis 3: Comparison: 68Ga-PSMA; PPV, composite standard, prostate or prostate bed: PPV of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy where available (composite standard of truth). In the prostate or prostate bed, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16; Sensitivity = 91.1, 95% CI 2-sided [86.2 to 100.00]
Statistical Analysis 4: Comparison: 68Ga-PSMA; Sensitivity, composite standard, prostate/prostate bed: We determined the sensitivity of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy (composite standard of truth). In the prostate or prostate bed, the sensitivity of conventional imaging ranges between 30-50%. The null hypothesis is that the sensitivity at 50% will be tested against the alternative hypothesis that the sensitivity is greater than 50%; Test type: Other — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16 Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); Sensitivity = 91.72, 95% CI 2-sided [86.74 to 100.00]
Statistical Analysis 5: Comparison: 68Ga-PSMA; PPV, composite standard, pelvic lymph nodes: PPV of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy where available (composite standard of truth). In the prostate or prostate bed, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%; Test type: Other — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16; PPV = 90.78, 95% CI 2-sided [85.74 to 100.00]
Statistical Analysis 6: Comparison: 68Ga-PSMA; Sensitivity, composite standard, pelvic lymph nodes: We determined the sensitivity of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy (composite standard of truth). In pelvic lymph nodes, the sensitivity of conventional imaging ranges between 30-50%. The null hypothesis is that the sensitivity at 50% will be tested against the alternative hypothesis that the sensitivity is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16; Sensitivity = 96.97, 95% CI 2-sided [93.20 to 100.00]
Statistical Analysis 7: Comparison: 68Ga-PSMA; PPV, composite standard, soft tissues: PPV of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy where available (composite standard of truth). In soft tissues, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.9e-15; PPV = 91.25, 95% CI 2-sided [84.19 to 100.00]
Statistical Analysis 8: Comparison: 68Ga-PSMA; Sensitivity, composite standard, soft tissues: We determined the sensitivity of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy (composite standard of truth). In soft tissues, the sensitivity of conventional imaging ranges between 30-50%. The null hypothesis is that the sensitivity at 50% will be tested against the alternative hypothesis that the sensitivity is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16; Sensitivity = 93.59, 95% CI 2-sided [86.99 to 100.00]
Statistical Analysis 9: Comparison: 68Ga-PSMA; PPV, composite standard, bone: PPV of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy where available (composite standard of truth). In bone tissues, the PPV of conventional imaging ranges between 30-50%. The null hypothesis is that the PPV at 50% will be tested against the alternative hypothesis that the PPV is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16; PPV = 95.17, 95% CI 2-sided [91.12 to 100.00]
Statistical Analysis 10: Comparison: 68Ga-PSMA; Sensitivity, composite standard, bone: We determined the sensitivity of 68Ga-PSMA-11 PET for presence of prostate cancer confirmed by conventional imaging, clinical follow-up, and histopathology/biopsy (composite standard of truth). In bone, the sensitivity of conventional imaging ranges between 30-50%. The null hypothesis is that the sensitivity at 50% will be tested against the alternative hypothesis that the sensitivity is greater than 50%; Test type: Superiority — Exact binomial proportion test, R statistical software package: R version 4.3.1 (2023-06-16); p < 0.0000001, Exact binomial proportion test — p-value = 2.2e-16; Sensitivity = 100, 95% CI 2-sided [97.85 to 100.00]

3. Secondary Outcome: Adverse Events of 68Ga-PSMA Administration
Description: The number of adverse events were determined through clinical assessment and categorized by CTCAE 4.0.
Time Frame: 24 - 72 hours post administration
Population: Participants in this arm were prostate cancer patients who experienced elevated PSA after definitive therapy with prostatectomy, radiation therapy (external beam or brachytherapy), or focal therapy of the prostate and received a 68Ga-PSMA-11 PET/CT scan.
Measure: Number; unit: events
Arm/Group | 68Ga-PSMA
Number analyzed (Participants) | 1181
events
  Serious adverse events | 1
  Adverse events | 2

4. Secondary Outcome: Detection Rates on a Per-patient Basis of 68Ga-PSMA-11 PET/CT
Description: Scan detection rates (in %) on a per-patient basis are given for specific PSA value ranges (a) 0.2<0.5, b) 0.5<1.0, c) 1.0<2.0, d) 2.0<5.0, e) >=5.0 ng/mL. Ideally, the 68Ga-PSMA-11 PET/CT scan detection rate would be 100% at any PSA range.
Time Frame: 12 months post scan
Population: Participants in this arm were prostate cancer patients who experienced elevated PSA after definitive therapy with prostatectomy, radiation therapy, or focal therapy of the prostate.
Measure: Number; unit: percentage of positive scans
Arm/Group | 68Ga-PSMA
Number analyzed (Participants) | 1181
percentage of positive scans
  PSA range 0.2 - < 0.5 ng/mL.: number analyzed (Participants) | 196
  PSA range 0.2 - < 0.5 ng/mL. | 55.1
  PSA range 0.5 - < 1.0 ng/mL.: number analyzed (Participants) | 170
  PSA range 0.5 - < 1.0 ng/mL. | 71.2
  PSA range 1.0 - < 2.0 ng/mL.: number analyzed (Participants) | 200
  PSA range 1.0 - < 2.0 ng/mL. | 85.5
  PSA range 2.0 - < 5.0 ng/mL.: number analyzed (Participants) | 265
  PSA range 2.0 - < 5.0 ng/mL. | 91.1
  PSA range 5.0 and above ng/mL.: number analyzed (Participants) | 350
  PSA range 5.0 and above ng/mL. | 95.4

5. Secondary Outcome: Impact of 68Ga-PSMA-11 PET on Clinical Management in BCR Patients
Description: The results of this outcome measure were evaluated using a treatment plan questionnaire given to the treating physician or practitioner before the scan, at approximately 1 month (2-30 days) after the 68Ga-PSMA-11 PET scan, and at approximately 6 months (range 3 - 12 months) after the 68Ga-PSMA-11 PET scan. The treatment plan questionnaire was provided with 11 choice options. Responses to the questionnaire were compared to determine whether physicians changed their treatment plans following the PET scan.
Time Frame: 2 days to 12 months following the scan.
Population: The intention was to count the number of prostate cancer patients and whether their treatment plans changed post scan based on physician survey responses and the participant's electronic medical record. Not all the physicians responded to surveys, and electronic records were not available for all participants, meaning data are missing for some patients.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Plans Up To 30 Days Post Scan: Treatment plan questionnaire given to the treating physician or practitioner at approximately 1 month (2-30 days) after the 68Ga-PSMA-11 PET scan.
- Treatment Plans At The End of the Study (One Year Post Scan): Final treatment plan based on surveys or the electronic medical record (obtained between 3 - 12 months after the 68Ga-PSMA-11 PET scan).
Arm/Group | Treatment Plans Up To 30 Days Post Scan | Treatment Plans At The End of the Study (One Year Post Scan)
Number analyzed (Participants) | 1181 | 1181
Participants
  Change in management from time before the scan | 886 | 374
  No change in management from time before the scan | 294 | 594
  Missing Data | 1 | 213

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events during and for 90 minutes after 68Ga-PSMA-11 administration. Patients were also contacted by phone to assess for the development of delayed adverse events up 3 days after 68Ga-PSMA-11 administration.
Description: Physicians received no intervention; therefore no adverse event data were collected.
Arm/Group | 68Ga-PSMA
All-Cause Mortality (participants affected / at risk) | 0/1181
Serious Adverse Events (participants affected / at risk) | 1/1181
Other Adverse Events (participants affected / at risk) | 2/1181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-PSMA (N=1181)
Coronary artery disease (Cardiac disorders) | 1 (1) — Subject with history of coronary artery disease and aortic stenosis developed chest pain during the research scan and was hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-PSMA (N=1181)
Dizziness (Cardiac disorders) | 1 (1) — Subject became dizzy and had balance problems following the research scan. Went to the emergency room and was further managed with medication.
Pain (General disorders) | 1 (1) — Patient developed pain due to positioning with his arms up during the imaging scan.

LIMITATIONS AND CAVEATS:
For Outcome Measure 5, a quality check was performed of the results by analyzing electronic medical records. The analysis showed the questionnaire responses about treatment plans collected post-scan did not align with the actual treatments listed in the medical records.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/74/NCT03396874/Prot_SAP_000.pdf